CLINICAL TRIAL: NCT06783127
Title: Clinical Outcomes of Use of Olaparib in Castration Resistant Prostate Cancer: An Observational Study
Brief Title: Clinical Outcomes of Use of Olaparib in Castration Resistant Prostate Cancer
Acronym: COROS
Status: Recruiting | Type: Observational
Sponsor: Santa Chiara Hospital (Other)
Responsible Party: Principal Investigator, Orazio Caffo, MD, Santa Chiara Hospital
Other Study IDs: A809
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer; Castrate Resistant Prostate Cancer; BRCA Mutation
MeSH Terms: conditions — Prostatic Neoplasms | interventions — olaparib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- mCRPC treated with olaparib: mCRPC patients who receive olaparib in daily clinical practice
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — Olaparib given according the clinical practice to BRCA positive mCRPC patients

SUMMARY:
This is an observational, retrospective/prospective, multicenter study designed to define, overall survival, clinical outcomes and predictive/prognostic factors of a consecutive population of mCRPC patients treated with olaparib in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

BRCA mutant Metastatic castration-resistant prostate cancer patients treatment with olaparib in clinical practice

Exclusion Criteria:

Olaparib treatment in a clinical trial

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: BRCA mutant Metastatic castration-resistant prostate cancer patients progressing after first-line ARPI who are treated with olaparib in clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
disease control | From the date of treatment start until the date of last follow-up or date of death from any cause, whichever came first, assessed up to 120 months
  projected survival from treatment start

SECONDARY OUTCOMES:
biochemical response | Through study completion, an average of 1 years
  rate of patients with PSA reduction > 50%
response rate | Through study completion, an average of 1 years
  rate of patients with measurable disease showing partial or complete response
PFS | From the date of treatment start until the date of first progression or date of death from any cause, whichever came first, assessed up to 120 months
  projected survival without progression
toxicity rate | Through study completion, an average of 1 years
  toxicity recorded during the treatment

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Sabrina Rossetti, Napoli
  - Orazio Caffo, Trento